CLINICAL TRIAL: NCT06995105
Title: Clinical Study to Evaluate the Safety and Efficacy of Personalized Tumor Neoantigen mRNA Therapy Combined With PD-1 Monoclonal Antibody and TACE for Advanced Hepatocellular Carcinoma
Brief Title: Personalized Tumor Neoantigen mRNA Therapy for Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, TingBo Liang, The chairman of the First Affiliated Hospital of Zhejiang University School of Medicine, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISLD-13
Record Dates: First submitted 2025-04-09; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (mRNA therapy+PD-1+anti-VEGFR+TACE) (Experimental): 1. After pathological diagnosis, the patient will pass the screening of the inclusion group and enter the study medication process;
  2. During the screening period, the patient can start TACE treatment first, and the subsequent treatment will be arranged by the researcher based on the patient's physical condition, disease progression, etc. The total number shall ≤ 4 times, and the interval between each two times shall be at least 4 weeks;
  3. After the patient enters the study medication process, he/she needs to first use sintilimab (200 mg) combined with bevacizumab (Dayoutong injection, 15 mg/kg), intravenous infusion, once every 3 weeks, until the patient is intolerant or the tumor progresses; the first use of sintilimab and Dayutong injection is the first day (D1)
  4. D43±3 (week 7±3 days), the first efficacy evaluation, if the patient has no disease progression, he/she will receive treatment (sintilimab Q3W + bevacizumab Q3W + the first batch of personalized mRNA inject Q3W)
  Interventions: Procedure: TACE; Drug: Sintilimab combined with Bevacizumab; Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection

INTERVENTIONS:
Procedure: TACE — The first day of TACE treatment is the first day (D1). TACE is started on D1. Subsequent TACE is arranged by the investigator based on a comprehensive assessment of the patient's physical condition, disease progression, adverse reactions, etc. The total number of TACEs shall not exceed 4 times, with at least 4 weeks between each two times.
Drug: Sintilimab combined with Bevacizumab — Sintilimab (200 mg) combined with bevacizumab (Dayoutong injection, 15 mg/kg), intravenous infusion, once every 3 weeks, until the patient is intolerant or the tumor progresses
Biological: individualized anti-tumor new antigen iNeo-Vac-R01 injection — The individualized anti-tumor new antigen iNeo-Vac-R01 injection was commissioned by Hangzhou Nuanjin Biotechnology Co., Ltd., and all patients were admitted into the therapeutic intervention group. According to the results of previous non-clinical studies, the individualized mRNA injection of 100 μ g was a tolerable dose.

SUMMARY:
This study is to evaluate the feasibility and safety of personalized tumor neoantigen mRNA therapy iNeo-Vac-R01 combined with PD-1 monoclonal antibody, anti-VEGFR monoclonal antibody and TACE regimen for the treatment of patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subjects who meet all the following inclusion criteria will enter the pre-screening stage of this study and undergo the lesion puncture process:

  1. Voluntarily sign the informed consent form;
  2. Aged ≥18 years and ≤75 years, regardless of gender;
  3. Strictly meet the 2018 American Association for Clinical Diagnosis of Liver Diseases (AASLD) clinical diagnostic criteria for HCC, and imaging assessment is unresectable/metastatic hepatocellular carcinoma (HCC), CNLC stage Ib to IIIb;
  4. Have not received systemic or local treatment for HCC in the past.
  5. According to the solid tumor efficacy evaluation criteria (RECIST 1.1), the investigators assess the presence of measurable lesions.
  6. Child-Pugh score within 7 points (including 7 points)
  7. Eastern Cooperative Oncology Group (ECOG) performance status score is 0 or 1;
  8. Adequate fresh tumor tissue samples can be obtained for exome and transcriptome sequencing analysis;
  9. The main organ functions of the heart, liver and kidney are normal:

     1. QTc (corrected QT interval) in the electrocardiogram: ≤450 milliseconds for men, or ≤470 milliseconds for women;
     2. Coagulation function: international normalized ratio (INR) ≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5 times ULN;
     3. Hematological indicators: white blood cells ≥3.5×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (HGB) ≥10 g/dL; platelet count (PLT) ≥80×109/L;
     4. Biochemical indicators: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (ALT or AST ≤ 5 times ULN is allowed for patients with liver metastasis and liver cancer); serum creatinine and urea nitrogen ≤ 1.5 times ULN;
  10. Male patients with fertility and female patients of childbearing age agree to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last administration of the trial drug; women of childbearing age include premenopausal women and women within 2 years after menopause;
  11. Able to follow the study protocol and follow-up process.

  (2) Subjects who meet all the following inclusion criteria will enter the formal screening phase of this study and enter the study medication process:
  1. Voluntarily sign the informed consent form;
  2. Aged ≥18 years and ≤75 years, regardless of gender;
  3. Primary hepatocellular carcinoma confirmed by pathology (histology or cytology);
  4. Have not received any systemic treatment.
  5. According to the solid tumor efficacy evaluation criteria (RECIST 1.1), the researcher assesses the presence of measurable lesions.
  6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
  7. Normal function of the heart, liver and kidney:

     1. QTc (corrected QT interval) in the electrocardiogram: ≤450 milliseconds for men, or ≤470 milliseconds for women;
     2. Coagulation function: international normalized ratio (INR) ≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5 times ULN;
     3. Hematological indicators: white blood cells ≥3.5×109/L; absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (HGB) ≥10 g/dL; platelet count (PLT) ≥80×109/L;
     4. Biochemical indicators: serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN (ALT or AST ≤ 5 times ULN is allowed for patients with liver metastasis and liver cancer); serum creatinine and urea nitrogen ≤ 1.5 times ULN;
  8. Male patients with fertility and female patients of childbearing age agree to take effective contraceptive measures from the signing of the informed consent form to 6 months after the last administration of the trial drug; women of childbearing age include premenopausal women and women within 2 years after menopause;
  9. Able to follow the study protocol and follow-up process.

     Exclusion Criteria:
* 1) Diffuse HCC. 2) Known fibrolamellar HCC, cholangiocarcinoma, and mixed HCC. 3) Concomitant tumor thrombus in the main portal vein or contralateral portal vein, superior mesenteric vein, or vena cava.

  4) History of meningeal disease; presence of central nervous system metastases or meningeal metastases.

  5) History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on screening chest CT.

  6) Patients with other malignant tumors at the same time, but basal cell carcinoma, thyroid cancer, cervical atypical hyperplasia, etc. that have been cured, have been in a disease-free state for more than 5 years or are considered by researchers to be less likely to relapse; 7) Patients with a history of bone marrow transplantation, allogeneic organ transplantation, or allogeneic hematopoietic stem cell transplantation; 8) Patients with immunosuppressants, that is, those who need to take immunosuppressants regularly 4 weeks before the screening period and during the clinical study, including but not limited to the following: those with severe asthma, autoimmune diseases or immunodeficiency, those who are treated with immunosuppressive drugs, and those with a known history of primary immunodeficiency; but excluding type 1 diabetes, autoimmune-related hypothyroidism requiring hormone treatment, and vitiligo and psoriasis that do not require systemic treatment; 9) Active bacterial or fungal infection confirmed by clinical diagnosis; active tuberculosis or history of tuberculosis; 10) Those with positive human immunodeficiency virus (HIV) antibody test, positive Treponema pallidum (TP) antibody test, active hepatitis C (positive hepatitis C virus (HCV) antibody and HCV RNA result is positive), active hepatitis B; 11) Herpes virus infection (except for those with scabs for more than 4 weeks); respiratory virus infection (except for those who have recovered for more than 4 weeks); 12) Uncontrolled complications include but are not limited to active infection, symptomatic congestive heart failure, unstable angina, arrhythmia; severe coronary artery disease or cerebrovascular disease, or other diseases that the investigators believe are not suitable for inclusion; 13) History of drug abuse, clinical, psychological or social factors that affect informed consent or research implementation; history of mental illness; 14) History of food, drug or vaccine allergy, or other potential immunotherapy allergies considered by the investigator.

  15) Pregnant or lactating women; 16) Those who the investigators believe are not suitable for inclusion or may not be able to complete this trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | The evaluation period was the dosing observation period and the safety follow-up period (21±3 days after the last dose).
  According to the Commonly Used Adverse Event Criteria (CTCAE version 5.0), the number of subjects with adverse events and/or dose-limiting toxicity was counted as an indicator of the safety and tolerable dose of iNeo-Vac-R01 injection.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
Disease control rate (DCR) | Up to 2 years
Conversion rate | Up to 2 years
  the proportion of patients with initially inoperable tumors who are successfully converted to patients who can undergo radical surgical resection after systemic treatment in conversion therapy
Progression-free survival （PFS） | Up to 2 years
Overall survival (OS) | Up to 2 years
Progression-free survival Rate（1-Y-PFS%, 2-Y-PFS%,3-Y-PFS%） | Up to 3 years
Overall Survival Rate (1-Y-OS%,2-Y-OS%,3-Y-OS%) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China